CLINICAL TRIAL: NCT04145674
Title: A Proof of Concept, Multicentre, Phase 2, Double-Blind, Randomized, Placebo-Controlled Study on the Efficacy, Safety and Tolerability of d-Methadone in Moderate to Very Severe Restless Legs Syndrome With Periodic Limb Movements: the Glu-REST Study
Brief Title: A Proof of Concept, Phase 2, Double-blind, Randomized Trial With d-Methadone Product Versus Placebo
Acronym: Glu-REST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mauro Manconi (Other)
Collaborators: Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor-Investigator, Mauro Manconi, Prof. MD, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSI-RLS-001
Record Dates: First submitted 2019-10-29; First posted 2019-10-30 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — D-methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25 mg d-methadone (Experimental): The experimental drug is a tablet formulation of d-methadone HCl in dose strength of 25 mg.
  Interventions: Drug: D-methadone
- Placebo (Placebo Comparator): The placebo is an exact match to the active tablets in size, color and marking without the active ingredient d-methadone HCl.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: D-methadone — Patients will take one tablet of 25 mg d-methadone once daily at 6 pm over a period of 30 days
  Other Names: esmethadone, dextromethadone, REL-1017
  Arms: 25 mg d-methadone
Other: Placebo — Patients will take one tablet of placebo once daily at 6 pm over a period of 30 days
  Arms: Placebo

SUMMARY:
Proof of concept, double-blind, randomized, placebo-controlled trial with d-methadone proposed for the first time for use in the treatment of patients diagnosed with primary, moderate to very severe Restless Legs Syndrome (RLS). Its glutamatergic mechanism of action might be effective on RLS arousal pattern and sleep disturbance which highly impair the quality of life of RLS's patients.

Patients will take the study drug/placebo once a day for 30 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary RLS.
* Moderate to very severe RLS defined as IRLS-RS score > 10.
* Written informed consent.
* Willingness and ability to participate in the trial

Exclusion Criteria:

* Positive history of known causes of secondary RLS.
* Any other concomitant treatment for RLS (wash-out period: at least 7 days).
* Moderate-severe sleep apnea defined as Apnea Hypopnea Index ≥ 15.
* History or presence of clinically significant abnormality as assessed by neurological examination which in the opinion of the Investigator would jeopardize the safety of the patients or the validity of the study results.
* Evidence of clinically significant hepatic or renal impairment
* History or family history of sudden unexplained death or long QT syndrome.
* Any 12-lead ECG with demonstration of QTc ≥ 450 msec or a QRS interval ≥ 120 msec at Screening.
* Concomitant use of psycho-drugs dopamine agonists and opioids (wash-out period: at least 7 days).
* History or presence of any condition in which an opioid is contraindicated
* History of allergy or hypersensitivity to methadone or related drugs.
* Any clinically significant neurological, sleep, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, chronic pain, psychiatric or gastrointestinal disorder.
* Women who are pregnant or breast feeding.
* Inability to follow the procedures of the study, (e.g. due to language problems, psychological disorders, dementia, etc. of the participant).
* Previous enrolment into the current study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-22 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of d-methadone | 30 days
  The percentage of responders to d-methadone treatment. A responder is defined as patient who has ≥ 50% reduction in the International RLS Rating Scale (IRLS-RS) score from baseline to end of the 30-day treatment period.

SECONDARY OUTCOMES:
Insomnia severity | 10 and 30 days
  Change in insomnia severity from baseline to the end of 10-day dosing period and to end of the treatment period assessed by a using the Insomnia Severity Index (ISI)
Change in Quality of life | 10 and 30 days
  Change in quality of life from baseline to the end of 10-day dosing period and to end of the treatment period assessed assessed by a using the Restless Legs Syndrome Quality of Life Questionnaire (RLSQoL)
Periodic limb movements of sleep index | 10 days
  Change in Periodic limb movements of sleep (PLMS) index from baseline to end of 10-day dosing period measured by means of polysomnography recording
Actigrafic parameters | 10 and 30 days
  Change from baseline to the end of 10-day dosing period and to end of the treatment period on Total Sleep Time, Sleep Latency and Sleep Efficacy acquired assessed by actigraphy with measurements performed one week prior to the start of treatment, during the 10-day dosing period and one week at the end of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Manconi, Prof. MD, Principal Investigator — Ente Ospedaliero Cantonale, Neurocenter of Southern Switzerland
Locations (4):
- Sleep Center, IRCCS San Raffaele, Milan, Italy
- Switzerland (3):
  - Schlaf-Wach-Epilepsie Zentrum, Inselspital, Bern
  - Neurologie / Schlaflabor Kantonsspital Graubünden, Chur
  - Sleep Center, Neurocenter of Southern Switzerland, Lugano

IPD SHARING:
Plan to Share IPD: Undecided